CLINICAL TRIAL: NCT06113315
Title: An Observational Study of Sarcoma Patients Treated With Immunotherapy at Memorial Sloan Kettering Cancer Center
Brief Title: A Study Involving Collection of Samples and Data From Sarcoma Patients Receiving Immunotherapy
Status: Enrolling by invitation | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 23-254
Record Dates: First submitted 2023-10-27; First posted 2023-11-02 (Actual); Last update posted 2025-10-27 (Actual); Status verified 2025-10

CONDITIONS: Sarcoma
Keywords: Immunotherapy; 23-254
MeSH Terms: conditions — Sarcoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Treatment-naïve patients who have not received any ICB and/or ACT treatment at time of consent: This is an observational prospective cohort study of patients with sarcoma treated with immune checkpoint blockade (ICB; anti-PD-1, PD-L1, and/or CTLA-4) or adoptive cell therapy (ACT; tumor infiltrating lymphocytes and/or engineered T cell receptor therapy) at Memorial Sloan Kettering Cancer Center (MSK).
- Treatment-experienced patients who have already received ICB and/or ACT treatment at time of consent: This is an observational prospective cohort study of patients with sarcoma treated with immune checkpoint blockade (ICB; anti-PD-1, PD-L1, and/or CTLA-4) or adoptive cell therapy (ACT; tumor infiltrating lymphocytes and/or engineered T cell receptor therapy) at Memorial Sloan Kettering Cancer Center (MSK).

SUMMARY:
The researchers are doing this study to improve their knowledge about immunotherapy use and how effective it is as a treatment for people with sarcoma by collecting information from participants' medical records who have been treated with immune checkpoint blockade or T-cell receptor-based therapy.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have a histologic diagnosis of sarcoma confirmed by an MSK pathologist.
* Any prospectively identified patient being treated or to be treated with an immune checkpoint inhibitor, such as anti-PD-1, anti-PD-L1, anti-CTLA-4, or anti-LAG3 inhibitor, either as monotherapy or in combination with additional systemic therapy OR any prospectively identified patient being treated or to be treated with ACT-based treatment including but not limited to lifileucil, Afamitresgene autoleucel, and letetresgene autoleuce o Novel immune checkpoints inhibitors that are developed after submission of this protocol will also be included) Please Note: there is no age requirement. Patients of all ages are eligible to enroll

Exclusion Criteria:

* Patient unwilling to consent to collection of historical and longitudinal clinicopathologic data in the patient medical record from baseline (the period prior to ICB or ACT initiation), during, and after ICB or ACT treatment

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All sarcoma patients who will undergo or are undergoing ICB-based or ACT-based treatment at MSK will be approached for participation in this observational study.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2023-10-27 (Actual); Primary Completion 2028-10 (Estimated); Study Completion 2028-10 (Estimated)

PRIMARY OUTCOMES:
prospectively collect and store blood | up to 5 years
  of sarcoma patients treated with ICB or ACT

CONTACTS AND LOCATIONS:
Overall Officials: Sandra D'Angelo, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (7):
- United States (7):
  - Memorial Sloan Kettering Cancer Center (All Protocol Activities), Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth (All Protocol Activities), Middletown, New Jersey
  - Memorial Sloan Kettering Bergen (All Protocol Activities), Montvale, New Jersey
  - Memorial Sloan Kettering Cancer Center Suffolk- Commack (All Protocol Activities), Commack, New York
  - Memorial Sloan Kettering Westchester (All Protocol Activities), Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering Nassau (All Protocol Activities), Uniondale, New York

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm